CLINICAL TRIAL: NCT03729882
Title: Prophylactic Endoscopic Ultrasound Gallbladder Drainage (EUS-GBD) in Patients With Unresectable Malignant Biliary Obstruction and Cystic Duct Orifice Involvement.
Brief Title: Primary EUS-GBD in Patients With Unresectable Malignant Biliary Obstruction and Cystic Duct Orifice Involvement.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Ecuatoriano de Enfermedades Digestivas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EUS-GBD
Record Dates: First submitted 2018-07-21; First posted 2018-11-05 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Acute Cholecystitis
Keywords: endoscopic ultrasound; acute cholecystitis; cholangiocarcinoma; gallbladder drainage; metallic stents
MeSH Terms: conditions — Cholecystitis, Acute; Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- EUS-guided gallbladder drainage (Other): In one arm, Endoscopic Ultrasound-Gallbladder Drainage (EUS-GBD) will be performed by using a 3,8 mm therapeutic echoendoscope and a lumen apposing metal stent ( Hot AXIOS™ Stent and Electrocautery Enhanced Delivered System; Boston Scientific Corporation, Natick, MA, USA) after conventional biliary drainage with self-expandable metallic stents during endoscopic retrograde cholangiopancreatography (ERCP).
  All procedures will be performed under general anesthesia.
  Interventions: Procedure: EUS-guided gallbladder drainage; Procedure: Non EUS-guided gallbladder drainage
- Non EUS-guided gallbladder drainage (Other): In the other arm, patients will undergo conventional biliary drainage with self-expandable metallic stent placement during ERCP evaluation without prophylactic EUS-GBD and will be considered as a Non EUS-guided gallbladder drainage.
  All procedures will be performed under general anesthesia.
  Interventions: Procedure: Non EUS-guided gallbladder drainage

INTERVENTIONS:
Procedure: EUS-guided gallbladder drainage — During ERCP evaluation a self-expandable metallic stent will be deployed in the common biliary duct of the patients enrolled in both arms of the present study. A prophylaxis gallbladder drainage will be done using a 3.8 mm working-channel linear-array therapeutic echoendoscope (EG3870UTK;Pentax, Hamburg, Germany) attached to an ultrasound console (Avius Hitachi, Tokyo, Japan) within a transgastric and/or transduodenal approaches to the gallbladder puncture followed by placement of a lumen apposing stent (LAMS) (AXIOS; Xlumena Inc, CA, USA) with a 10 mm luminal diameter and a dumbbell-shaped flanges to bring together the 2 walls in apposition. These feature of the Axios decrease the risk for bile leak, stent migration, and stent occlusion.
  Arms: EUS-guided gallbladder drainage
Procedure: Non EUS-guided gallbladder drainage — During ERCP evaluation a self-expandable metallic stent will be deployed in the common biliary duct of the patients enrolled in both arms of the present study. If the patient had an acute cholecystitis will be sent to surgery and be considered as a Non EUS-guided gallbladder drainage

SUMMARY:
to determine if primary prophylaxis with Endoscopic Ultrasound-Gallbladder Drainage (EUS-GBD) in unresectable cancer patients with the orifice of the cystic duct (OCD) involvement is superior to conservative management (Non EUS-guided gallbladder drainage).

DETAILED DESCRIPTION:
Endoscopic biliary drainage with a self-expandable metal stent (SEMS) is an accepted form of palliative therapy for distal malignant biliary obstruction (MBO); it is a low invasive procedure with a long-term patency.

Covered SEMSs have a longer patency than uncovered SEMSs in patients with MBO, because covered SEMSs can prevent tumor ingrowth. However, complications of covered SEMSs include stent occlusion, migration, kinking, non-occlusion cholangitis, liver abscess, pancreatitis and cholecystitis.

Nonsurgical decompression of the gallbladder is urgently needs to prevent sepsis, perforation and death in patients with acute cholecystitis. Several risk factors of cholecystitis after SEMS placement for distal MBO have been reported: however, tumor involvement to the orifice of the cystic duct (OCD) is the major predictive factor for cholecystitis after endoscopic SEMSs placement for distal MBO palliative treatment .

Acute cholecystitis related to SEMSs deployment was evaluated in 2009, by using endoscopic trans-papillary gallbladder drainage (TPGBD) in 11 individuals in whom SEMSs covered the OCD. None episode of cholecystitis was reported, however TPGBD is a difficult technique with a high rate of stent dislodgement and reintervention needed.

EUS-GBD by using a lumen apposing metal stent have been proposed, but only for acute cholecystitis treatment or symptomatic gallbladder hydrops, never as a prophylactic technique.

The aim of this study if to determine if primary prophylaxis EUS-GBD in patients with distal malignant biliary obstruction and the OCD involvement is superior than conservative management. Also, a cost-effectiveness analysis will be done in both arm groups.

This would be the first trial to study the effect of prophylactic EUS-GBD prior SEMSs deployment in patients with distal malignant biliary obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old.
* Obtained written consent for procedures
* Unresectable malignant biliary obstruction diagnosed by Endoscopic Ultrasound and confirmed by confocal laser endomicroscopy (CLE) during cholangioscopy and histopathology.
* Tumor involvement to the orifice of the cystic duct.
* Self-expandable metallic plastic stent deployment as palliative therapy for distal biliary obstruction.

Exclusion Criteria:

* Under 18 years old.
* Refuse to sign written informed consent.
* Pregnancy
* Previous cholecystectomy
* Acute cholecystitis prior enrollment
* Severe ascites that increases the distance between gastric or duodenal and gallbladder walls.
* Large vessel between the gallbladder and gastric-duodenal wall.
* Coagulopathy
* Intrahepatic cholangiocarcinoma
* Previous gallbladder drainage by percutaneous or endoscopic techniques.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2020-07-27 (Actual)

PRIMARY OUTCOMES:
Ocurrence of acute cholecystitis | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  • Occurrence of acute cholecystitis according to Tokyo guidelines 2013: Clinical symptoms showing right upper or epigastric pain or tenderness, signs of systematic inflammation (fever, elevated white blood cell count, and C-reactive protein), or positive findings on abdominal ultrasonography (US) or computed tomography (CT).

SECONDARY OUTCOMES:
Technical success rate: EUS-GBD | from the beginning of the EUS-GBD procedure and 10 minutes after LAMS placement.
  as the ability of access and drain the gallbladder by placement of a drainage stent: lumen apposing metal stent ( Hot AXIOS™ Stent and Electrocautery Enhanced Delivered System; Boston Scientific Corporation, Natick, MA, USA).
Clinical success rate: | since enrollment until 30-days follow up.
  non-occurrence of acute cholecystitis during follow up OR successful SEMS placement with biliary decompression and relief of jaundice pruritus.
adverse events | from the beginning of the procedure until 30 days.
  any procedure-related adverse event (anesthesia, EUS-GBD, ERCP).
presence of pus during EUS-GBD | immediate after EUS-GBD.
  endoscopic visualization of pus after EUS-GBD. Yes or no.
Duration of the lumen apposing stent patency in the EUS-GBD arm study | the interval (days) between the time of stent placement and that of stent malfunction or patient death, whichever came first, assessed up to 12 months.
  Duration of the lumen apposing stent patency in the EUS-GBD arm study
Need for gallbladder re-intervention. | from the end of the procedure until the date of first documented episode of acute cholecystitis through 12 months follow-up
  on EUS-GBD patients arm, need for a new gallbladder drainage (surgical or percutaneous) due to the occurrence of acute cholecystitis.
Total length of hospital stay | from the beginning of hospitalization until discharge date or death since enrollment through 12 months follow-up
  it will be measured on both arms study when patients require hospitalization due to any procedure adverse event, cholecystitis and related procedures (cholecystectomy, percutaneous drainage)
Total health-care related cost of both arm participants. | from the end of conventional biliary drainage until the date of 12 months follow-up.
  total health-are related cost in all participants from each arm.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Robles-Medranda, Principal Investigator — Instituto Ecuatoriano de Enfermedades Digestivas
Locations (1):
- Instituto Ecuatoriano de Enfermedades Digestivas, Guayaquil, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gosain S, Bonatti H, Smith L, Rehan ME, Brock A, Mahajan A, Phillips M, Ho HC, Ellen K, Shami VM, Kahaleh M. Gallbladder stent placement for prevention of cholecystitis in patients receiving covered metal stent for malignant obstructive jaundice: a feasibility study. Dig Dis Sci. 2010 Aug;55(8):2406-11. doi: 10.1007/s10620-009-1024-9. Epub 2009 Nov 4. PMID 19888656
- [Background] Nakai Y, Isayama H, Kawakubo K, Kogure H, Hamada T, Togawa O, Ito Y, Matsubara S, Arizumi T, Yagioka H, Takahara N, Uchino R, Mizuno S, Miyabayashi K, Yamamoto K, Sasaki T, Yamamoto N, Hirano K, Tada M, Koike K. Metallic stent with high axial force as a risk factor for cholecystitis in distal malignant biliary obstruction. J Gastroenterol Hepatol. 2014;29(7):1557-62. doi: 10.1111/jgh.12582. PMID 24628054
- [Background] Isayama H, Kawabe T, Nakai Y, Tsujino T, Sasahira N, Yamamoto N, Arizumi T, Togawa O, Matsubara S, Ito Y, Sasaki T, Hirano K, Toda N, Komatsu Y, Tada M, Yoshida H, Omata M. Cholecystitis after metallic stent placement in patients with malignant distal biliary obstruction. Clin Gastroenterol Hepatol. 2006 Sep;4(9):1148-53. doi: 10.1016/j.cgh.2006.06.004. Epub 2006 Aug 14. PMID 16904950
- [Background] Shimizu S, Naitoh I, Nakazawa T, Hayashi K, Miyabe K, Kondo H, Yoshida M, Yamashita H, Umemura S, Hori Y, Ohara H, Joh T. Predictive factors for pancreatitis and cholecystitis in endoscopic covered metal stenting for distal malignant biliary obstruction. J Gastroenterol Hepatol. 2013 Jan;28(1):68-72. doi: 10.1111/j.1440-1746.2012.07283.x. PMID 23020651
- [Background] Xu MM, Kahaleh M. EUS-guided transmural gallbladder drainage: a new era has begun. Therap Adv Gastroenterol. 2016 Mar;9(2):138-40. doi: 10.1177/1756283X15618178. No abstract available. PMID 26929775
- [Background] Irani S, Ngamruengphong S, Teoh A, Will U, Nieto J, Abu Dayyeh BK, Gan SI, Larsen M, Yip HC, Topazian MD, Levy MJ, Thompson CC, Storm AC, Hajiyeva G, Ismail A, Chen YI, Bukhari M, Chavez YH, Kumbhari V, Khashab MA. Similar Efficacies of Endoscopic Ultrasound Gallbladder Drainage With a Lumen-Apposing Metal Stent Versus Percutaneous Transhepatic Gallbladder Drainage for Acute Cholecystitis. Clin Gastroenterol Hepatol. 2017 May;15(5):738-745. doi: 10.1016/j.cgh.2016.12.021. Epub 2016 Dec 30. PMID 28043931
- [Background] Hatanaka T, Itoi T, Ijima M, Matsui A, Kurihara E, Okuno N, Kobatake T, Kakizaki S, Yamada M. Efficacy and Safety of Endoscopic Gallbladder Stenting for Acute Cholecystitis in Patients with Concomitant Unresectable Cancer. Intern Med. 2016;55(11):1411-7. doi: 10.2169/internalmedicine.55.5820. Epub 2016 Jun 1. PMID 27250045
- [Background] Choi JH, Kim HW, Lee JC, Paik KH, Seong NJ, Yoon CJ, Hwang JH, Kim J. Percutaneous transhepatic versus EUS-guided gallbladder drainage for malignant cystic duct obstruction. Gastrointest Endosc. 2017 Feb;85(2):357-364. doi: 10.1016/j.gie.2016.07.067. Epub 2016 Aug 24. PMID 27566055
- [Background] Dollhopf M, Larghi A, Will U, Rimbas M, Anderloni A, Sanchez-Yague A, Teoh AYB, Kunda R. EUS-guided gallbladder drainage in patients with acute cholecystitis and high surgical risk using an electrocautery-enhanced lumen-apposing metal stent device. Gastrointest Endosc. 2017 Oct;86(4):636-643. doi: 10.1016/j.gie.2017.02.027. Epub 2017 Mar 1. PMID 28259594